CLINICAL TRIAL: NCT04187898
Title: Open-Label, Phase 1 Study to Evaluate Duration of Severe Neutropenia After the Same-Day, Varying Dosing Time Schedules of Eflapegrastim Administration in Patients With Breast-Cancer Receiving Docetaxel and Cyclophosphamide
Brief Title: Open-Label, Phase 1 Study to Evaluate Duration of Severe Neutropenia After Same-Day Dosing of Eflapegrastim in Patients With Breast-Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Spectrum Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SPI-GCF-104
Record Dates: First submitted 2019-10-30; First posted 2019-12-05 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Neutropenia; Breast Cancer
Keywords: Neutropenia; Early Stage Breast Cancer; Long-acting Myeloid Growth Factor; Docetaxel + Cyclophosphamide (TC) Chemotherapy
MeSH Terms: conditions — Neutropenia; Breast Neoplasms | interventions — eflapegrastim; Docetaxel; Cyclophosphamide

STUDY DESIGN:
Intervention Model Description: Considering two-phase study, where Expansion Phase followed Early Phase. The dosing within the Early Phase was in parallel assignment wherein participants were assigned to three arms in a 1:1:1 ratio. Patients completing Early Phase will enter the Expansion Phase to receive dosing in a single arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Early Phase: Eflapegrastim @ 30mins post TC (Experimental): Eflapegrastim (13.2 mg/0.6 mL fixed dose, equivalent to 3.6 mg granulocyte colony-stimulating factor [G-CSF]).
  Supplied in prefilled single-use syringes for subcutaneous injection.
  Cycle 1: Administered on the same day as TC chemotherapy, 30 minutes from the end of TC administration.
  Cycles 2-4: Administered 24 hours after TC chemotherapy administration.
  Each cycle is 21 days.
  Interventions: Biological: Eflapegrastim; Drug: Docetaxel; Drug: Cyclophosphamide
- Early Phase: Eflapegrastim @ 3 hours post TC (Experimental): Eflapegrastim (13.2 mg/0.6 mL fixed dose, equivalent to 3.6 mg G-CSF).
  Supplied in prefilled single-use syringes for subcutaneous injection.
  Cycle 1: Administered on the same day as TC chemotherapy, 3 hours from the end of TC administration.
  Cycles 2-4: Administered 24 hours after TC chemotherapy administration.
  Each cycle is 21 days.
  Interventions: Biological: Eflapegrastim; Drug: Docetaxel; Drug: Cyclophosphamide
- Early Phase: Eflapegrastim @ 5 hours post TC (Experimental): Eflapegrastim (13.2 mg/0.6 mL fixed dose, equivalent to 3.6 mg G-CSF).
  Supplied in prefilled single-use syringes for subcutaneous injection.
  Cycle 1: Administered on the same day as TC chemotherapy, 5 hours from the end of TC administration.
  Cycles 2-4: Administered 24 hours after TC chemotherapy administration.
  Each cycle is 21 days.
  Interventions: Biological: Eflapegrastim; Drug: Docetaxel; Drug: Cyclophosphamide
- Expansion Phase: Eflapegrastim @ 30 mins post TC (Experimental): Eflapegrastim (13.2 mg/0.6 mL fixed dose, equivalent to 3.6 mg G-CSF).
  Supplied in prefilled single-use syringes for subcutaneous injection.
  Cycles 1-4: Administered on the same day as TC chemotherapy, 30 minutes following the end of TC administration.
  Each cycle is 21 days.
  Interventions: Biological: Eflapegrastim; Drug: Docetaxel; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: Eflapegrastim — Administered in Cycle 1, 30 minutes after TC chemotherapy.
  Administered in Cycles 2-4, on day 2 of each cycle.
  Arms: Early Phase: Eflapegrastim @ 30mins post TC
Biological: Eflapegrastim — Administered in Cycle 1, 3 hours after TC chemotherapy.
  Administered in Cycles 2-4, on day 2 of each cycle.
  Arms: Early Phase: Eflapegrastim @ 3 hours post TC
Biological: Eflapegrastim — Administered in Cycle 1, 5 hours after TC chemotherapy.
  Administered in Cycles 2-4, on day 2 of each cycle.
  Arms: Early Phase: Eflapegrastim @ 5 hours post TC
Biological: Eflapegrastim — Administered in Cycles 1-4, 30 mins after TC chemotherapy.
  Arms: Expansion Phase: Eflapegrastim @ 30 mins post TC
Drug: Docetaxel — 75 mg/m^2 IV infusion.
  Administered on Day 1 of each cycle.
  Other Names: Taxotere
Drug: Cyclophosphamide — 600 mg/m^2 IV infusion.
  Administered on Day 1 of each cycle.
  Other Names: Cytoxan

SUMMARY:
The purpose of this study is to compare the effect of Eflapegrastim on duration of neutropenia in patients with early-stage breast cancer when administered at varying intervals following Docetaxel and Cyclophosphamide administration.

DETAILED DESCRIPTION:
This is a Phase 1, randomized, open label, actively-controlled study to evaluate the same day dosing of Eflapegrastim on duration of neutropenia when administered at varying intervals following Docetaxel and Cyclophosphamide (TC) chemotherapy in patients with early-stage breast cancer.

The study will be conducted in two phases: Early Phase and Expansion Phase.

1. In the Early Phase, approximately 45 patients were enrolled and randomized in a 1:1:1 ratio to 3 dosing time schedule arms. Each cycle was of 21 days. Total 4 cycles were evaluated for this phase. On Day 1 of Cycle 1, patients received Docetaxel and Cyclophosphamide (TC) chemotherapy followed by administration of Eflapegrastim at 1 of 3-time schedules post-TC (30 minutes [mins], 3 hours or 5 hours). During Cycles 2-4, patients received Eflapegrastim 24 hours after TC administration (on Day 2).
2. In the Expansion Phase, additional 45 patients will be enrolled in Cycles 1-4, who will receive fixed dose of Eflapegrastim 30 mins after TC administration (on Day 1).

Safety evaluations will be conducted once the first 3 patients (for Early Phase) and the first 6 patients (for Expansion Phase) have completed Cycle 1 to determine if it is safe for patients to continue in that particular treatment arm.

ELIGIBILITY:
Inclusion Criteria:

* Willing and capable of giving written Informed Consent and able to adhere to study drug dosing time and blood draw schedules
* New diagnosis of histologically confirmed early-stage breast cancer (ESBC), defined as operable Stage I to Stage IIIA breast cancer
* Candidate to receive adjuvant or neoadjuvant TC chemotherapy
* Age must be at least 18 years for the Early Phase, and between 18 to ≤55 years for the Expansion Phase
* ANC ≥1.5×10^9/liter (L).
* Platelet count ≥100×10^9/liter (L).
* Hemoglobin >10 grams per deciliter (g/dL).
* Calculated creatinine clearance >50 milliliter per minute (mL/min).
* Total bilirubin ≤1.5 milligrams per deciliter (mg/dL).
* Aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase (SGOT) and alanine aminotransferase (ALT)/serum glutamic pyruvic transaminase (SGPT) ≤2.5×upper limit of normal (ULN).
* Alkaline phosphatase ≤2.0×ULN.
* Eastern Cooperative Oncology Group (ECOG) ≤2
* Willing to practice 2 forms of contraceptives (1 must be a barrier method), from study entry through 30 days after last dose of study drug/ early discontinuation
* Negative urine pregnancy test within 30 days before randomization

Exclusion Criteria:

* Active concurrent malignancy (except non melanoma skin cancer or carcinoma in situ of the cervix) or life-threatening disease
* Known sensitivity to Escherichia coli (E. coli) derived products
* Concurrent adjuvant cancer therapy other than the trial-specified therapies
* Locally recurrent/metastatic breast cancer
* Previous exposure to filgrastim, pegfilgrastim, or other G-CSF products in clinical development within 3 months prior to the administration of study drug
* Receiving anti-infectives, has an underlying medical condition or other serious illness that would impair the ability to receive protocol-specified treatment
* Used any investigational drugs, biologics, or devices within 30 days prior to study treatment or plans to use any of these during the course of the study
* Prior bone marrow or stem cell transplant
* Prior radiation therapy within 30 days prior to enrollment
* Major surgery within 30 days prior to enrollment
* Pregnant or breastfeeding

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2020-03-11 (Actual); Primary Completion 2024-07-16 (Actual); Study Completion 2024-08-16 (Actual)

PRIMARY OUTCOMES:
Time to Recovery of Absolute Neutrophil Count (ANC) From Nadir to ≥1.5×10^9/L in Cycle 1 | Cycle 1 is 21 days
  Time to ANC Recovery is defined as the time from chemotherapy administration until the patient's ANC increases to ≥1.5×10^9/liter (L) after the expected nadir.

SECONDARY OUTCOMES:
Duration of Grade 4 Neutropenia (DSN) in Cycle 1 | Cycle 1 is 21 days
  DSN is defined as the number of days of severe neutropenia where the ANC<0.5x10^9/L from the first occurrence of an ANC below the threshold.
Proportion of Patients With Grade 4 Neutropenia in Cycle 1 | Cycle 1 is 21 days
Incidence of Grade 3 Febrile Neutropenia (FN) in Cycle 1 | Cycle 1 is 21 days
  FN is defined as having an ANC<1.0x10^9/L and either a single temperature of >38.3 degrees Celsius (101.0 Fahrenheit [F]) or a sustained temperature of >38.0 degrees Celsius (100.4 F).
Incidence of Neutropenic Complications, Including Hospitalization due to Neutropenia, FN, and use of Anti-infectives During Cycle 1 | Cycle 1 is 21 days
Expansion Phase: Time to Recovery of ANC From Nadir to ≥1.5×10^9/L in Cycles 2-4 | Cycles 2-4 (cycle length=21 days) (up to approximately 63 days)
  Time to ANC Recovery is defined as the time from chemotherapy administration until the patient's ANC increases to ≥1.5×10^9/L after the expected nadir.
Expansion Phase: DSN in Cycles 2-4 | Cycles 2-4 (cycle length=21 days) (up to approximately 63 days)
  DSN is defined as the number of days of severe neutropenia where the ANC <0.5x10^9/L from the first occurrence of an ANC below the threshold.
Expansion Phase: Proportion of Patients With Grade 4 Neutropenia in Cycles 2-4 | Cycles 2-4 (cycle length=21 days) (up to approximately 63 days)
Expansion Phase: Incidence of FN in Cycles 2-4 | Cycles 2-4 (cycle length=21 days) (up to approximately 63 days)
  FN is defined as having an ANC<1.0x10^9/L and either a single temperature of >38.3 degrees Celsius (101.0 F) or a sustained temperature of >38.0 degrees Celsius (100.4 F).
Expansion Phase: Incidence of Neutropenic Complications, Including Hospitalization due to Neutropenia, FN, and use of Anti-infectives During Cycles 2-4 | Cycles 2-4 (cycle length=21 days) (up to approximately 63 days)
Number of Patients With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) as a Measure of Safety | Up to approximately 40 days after the last dose of study treatment or early study discontinuation (up to approximately 4 months)
Proportion of Patients Discontinuing Because of a TEAE | Up to approximately 40 days after the last dose of study treatment or early study discontinuation (up to approximately 4 months)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - ACRC/ Arizona Clinical Research Center, Tucson, Arizona
  - Yuma Regional Medical Center Cancer Center, Yuma, Arizona
  - Pacific Cancer Medical Center, Anaheim, California
  - City of Hope, Long Beach, California
  - BRCR Medical Center, Inc., Plantation, Florida
  - Bond & Steele Clinic, P.A., Winter Haven, Florida
  - SCL Health Research Institute, Inc., Billings, Montana
  - Mercy Health Youngstown, Youngstown, Ohio

IPD SHARING:
Plan to Share IPD: No